CLINICAL TRIAL: NCT01822405
Title: Treatment of Radiation-induced Fibrosis in the Upper Aerodigestive Tract Cancer by a Combination of Pentoxifylline-tocopherol and Hyperbaric Oxygen
Acronym: ORT-OXI-2009
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario de Canarias (Other)
Collaborators: Instituto Médico Tinerfeño IMETISA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORT-OXI-2009
Record Dates: First submitted 2013-03-21; First posted 2013-04-02 (Estimated); Last update posted 2013-04-02 (Estimated); Status verified 2013-03

CONDITIONS: Fibrosis
MeSH Terms: conditions — Fibrosis | interventions — Pentoxifylline; Tocopherols; Hyperbaric Oxygenation

ARMS (2):
- Pentoxifylline + Tocopherol (Active Comparator): Pentoxifylline 800 mg/day (400 mg/12hours) + Tocopherol 1000 mg/day oral during 6 months
  Interventions: Drug: pentoxifylline with tocopherol
- pentoxifylline + tocopherol + Hyperbaric Oxygen Therapy (Experimental)
  Interventions: Other: pentoxifylline+tocopherol + Hyperbaric Oxygen Therapy

INTERVENTIONS:
Drug: pentoxifylline with tocopherol — Pentoxifylline 800 mg/day (400 mg/12hours) + Vitamin E (alfa-tocopherol) 1000 mg/day,oral during 6 months
  Arms: Pentoxifylline + Tocopherol
Other: pentoxifylline+tocopherol + Hyperbaric Oxygen Therapy — pentoxifylline 800 mg/day (400 mg/12hours) + Vitamin E (alfa-tocopherol) 1000 mg/day, oral during 6 months.
  Hyperbaric Oxygen Therapy at 100% in 25 sessions of 90 minutes 5 days per week (5 weeks) at 2,4 Ata in Hyperbaric chamber, starting in 3 or 9 weeks after randomization and beginning of drug treatment.
  Arms: pentoxifylline + tocopherol + Hyperbaric Oxygen Therapy

SUMMARY:
The pentoxifylline used with tocopherol achieves a certain effectiveness in the treatment of the fibrosis.

Hyperbaric oxygen therapy has been recommended and used in a wide variety of medical conditions including the treatment of delayed radiation injuries (soft tissue and bony radiation necrosis). The hyperbaric oxygen therapy increases the formation of granulation tissue and produces angiogenesis maintained after use.

DETAILED DESCRIPTION:
Patients with head and neck tumors often present superficial radiation induced fibrosis and other late complications of radiotherapy that can seriously affect their quality of life.

The pentoxifylline used with tocopherol achieves a certain effectiveness in the treatment of the fibrosis.

Hyperbaric oxygen therapy has been recommended and used in a wide variety of medical conditions including the treatment of delayed radiation injuries (soft tissue and bony radiation necrosis). The hyperbaric oxygen therapy increases the formation of granulation tissue and produces angiogenesis maintained after use.

Both treatments in combination could produce a synergistic effect because the angiogenesis induced by hyperbaric oxygen therapy allow better access to drugs to the injury. The magnetic resonance, provides data of the fibrosis and other side effects of radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years and under 70 years old.
2. Patients who have received radiotherapy after being diagnosed with cancer of upper aerodigestive tract, and have skin toxicity grade II or higher.
3. Follow-up for at least a year after the radiation treatment is completed.
4. Absence of tumor at the time of recruitment.
5. Patients with the capacity to give informed consent

Exclusion Criteria:

1. Allergy or hypersensitivity to Pentoxifylline or others xanthines, or to Tocopherol (vitamin E).
2. Patients taking oral anticoagulants (acenocoumarol, warfarin).
3. Known hemorrhagic/coagulation disorder.
4. Vitamin K deficiency due to any cause.
5. Use of estrogens oral contraceptives.
6. Serious bleeding or extensive retinal hemorrhage.
7. Ischaemic heart diseases, including recent Myocardial Infarction.
8. Serious cardiac arrhythmia.
9. Severe liver disease.
10. Severe renal failure (creatinine clearance <30 mL/min).
11. Hypotension.
12. Patients with metal objects or electronic devices such as cardiac pacemakers, artificial heart valves or cochlear implants, or any other contraindication for MRI
13. Contraindication for Hyperbaric oxygen therapy.
14. Patients with mobility problems.
15. Female patients who are pregnant or lactating
16. Any other situation or condition that, in the opinion of the investigator, may interfere with optimal participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2010-07; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Change in skin fibrosis measured by MRI | From baseline to 6 month of starting treatment
  The change is calculated as the latest time point (6 months) minus the earliest time point (baseline)

SECONDARY OUTCOMES:
Clinical assessment of the radiation late (delayed) toxicity for mucosal membranes, salivary glands, larynx and skin by the LENT-SOMA scale (Late Effect Normal Tissue Task Force / Subjective, Objective, Management, Analytic scale) | Baseline and 6 months
  The change is calculated as the latest time point (6 months) minus the earliest time point (baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Otón, MD, Principal Investigator — Hospital Universitario de Canarias
Locations (1):
- Hospital Universitario de Canarias, San Cristóbal de La Laguna, S/C de Tenerife, Spain